CLINICAL TRIAL: NCT02896023
Title: Sonographic and Laboratory Predictors of Ovarian Reserve in Infertile Women
Brief Title: Predictors of Ovarian Reserve in Infertile Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 154
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Reserve
Keywords: predictors; ovarian reserve; infertile women
MeSH Terms: interventions — Menotropins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregnant (Active Comparator): women with positive pregnancy test after induction of ovulation and ICSI
  Interventions: Drug: human menopausal gonadotropin
- Not pregnant (Active Comparator): women with negative pregnancy test after induction of ovulation and ICSI
  Interventions: Drug: human menopausal gonadotropin

INTERVENTIONS:
Drug: human menopausal gonadotropin — Induction of ovulation followed by ICSI
  Other Names: menogon

SUMMARY:
Patients will be subjected to:

A. Clinical evaluation including history and examination

B. Ultrasonographic evaluation of Ovarian Morphometry:

* Patients will be evaluated in early follicular phase of the menstrual flow (cycle's days 1-3) by TVS scanning; using MINDRAY DP-1100 Plus Digital Machine, 7.5MHz, China, by only one examiner to avoid inter-observer variations.
* Ovarian images will be procured in the sagittal and coronal planes and the frozen image reflecting the largest ovarian dimensions will be utilized for the measurement of ovarian length, width, and height (cm) as per standard clinical practice. Mean values of both ovaries will be used. Ovarian volume will be calculated from ellipsoid volume formula, {Ovarian volume = Ovarian Width (D1) × Ovarian Length (D2) ×Ovarian Height (D3) × 0 .523}
* Antral follicle count will be determined for each patient

C. Laboratory Evaluation:

Blood samples will be collected in the early follicular phase. Samples will be immediately centrifuged and serum saved at -20 degrees for measurement of:

* Anti Mullerian Hormone (AMH)
* Follicle Stimulating Hormone (FSH)
* Estradiol (E2) Using electro-chemiluminescence immunoassay (ELICA)

DETAILED DESCRIPTION:
Patients will be subjected to:

A. Clinical evaluation including history and examination

B. Ultrasonographic evaluation of Ovarian Morphometry:

* Patients will be evaluated in early follicular phase of the menstrual flow (cycle's days 1-3) by TVS scanning; using MINDRAY DP-1100 Plus Digital Machine, 7.5MHz, China, by only one examiner to avoid inter-observer variations.
* Ovarian images will be procured in the sagittal and coronal planes and the frozen image reflecting the largest ovarian dimensions will be utilized for the measurement of ovarian length, width, and height (cm) as per standard clinical practice. Mean values of both ovaries will be used. Ovarian volume will be calculated from ellipsoid volume formula, {Ovarian volume = Ovarian Width (D1) × Ovarian Length (D2) ×Ovarian Height (D3) × 0 .523}
* Antral follicle count will be determined for each patient

C. Laboratory Evaluation:

Blood samples will be collected in the early follicular phase. Samples will be immediately centrifuged and serum saved at -20 degrees for measurement of:

* Anti Mullerian Hormone (AMH)
* Follicle Stimulating Hormone (FSH)
* Estradiol (E2) Using electro-chemiluminescence immunoassay (ELICA)

ELIGIBILITY:
Inclusion Criteria:

* less than 39 years old,
* normal menstrual cycle with a range of 24 to 35 days
* normal seum prolactin.
* normal uterine cavity determined by previous hysterosalpingography or hysteroscopy

Exclusion Criteria:

* smokers
* endometriosis
* Women with endometriosis;
* abnormal endocrine functions such as diabetes mellitus, thyroid disorders, and adrenal abnormalities; general diseases, those with ovarian cysts, or those who have azospermia partners.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
positive pregnancy test | 14 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes